CLINICAL TRIAL: NCT03242512
Title: Phase I Trial of Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Fully Human Monoclonal Antibody to RANKL (TK006) in Post-menopausal Women.
Brief Title: Assessment of Anti-RANKL Antibody in Post-menopausal Women
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu T-Mab Biopharma Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TK006-101
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Osteoporosis
Keywords: RANKL; osteoporosis; bone resorption; post-menopausal women; TK006
MeSH Terms: conditions — Osteoporosis; Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30 mg single dose cohort (Experimental): Subjects would receive a 30 mg single dose of TK006.
  Interventions: Biological: TK006
- 60 mg single dose cohort (Experimental): Subjects would receive a 60 mg single dose of TK006.
  Interventions: Biological: TK006
- 120 mg single dose cohort (Experimental): Subjects would receive a 120 mg single dose of TK006.
  Interventions: Biological: TK006

INTERVENTIONS:
Biological: TK006 — Subcutaneous injection
  Other Names: fully human monoclonal anti-RANKL antibody

SUMMARY:
This is a single-center, open-label, dose-escalating study to evaluate the safety, pharmacokinetics, immunogenicity, and preliminary efficacy of single dose subcutaneous injection of a fully human monoclonal antibody of receptor activator for nuclear factor-κ B ligand (RNAKL) (code name: TK006) in postmenopausal women.

DETAILED DESCRIPTION:
This is a phase I, open-label, single-dose, dose escalation study in postmenopausal women conducted at single center.

The objectives are to assess the safety and tolerability, effects on bone turnover measured by biochemical markers and bone density, and the pharmacokinetics and immunogenicity of a fully human monoclonal antibody of receptor activator for nuclear factor-κ B ligand (RNAKL), (code name: TK006).

Subjects would sequentially enroll in one of three cohorts. Subjects in the first cohort would receive a single 30-mg subcutaneous injection of TK006. If no safety signals are observed in the first cohort after 28 days, subjects would enroll in the second cohort and receive a single 60-mg subcutaneous injection of TK006. After an 28-day period for observation of safety of the second dose, subjects would enroll in the third cohort and receive a single 120-mg subcutaneous injection of TK006.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who provide informed consent voluntarily;
2. Women who are postmenopausal defined as being amenorrheic for at least 24-month, and follicule-stimulating hormone (FSH)>40 U/L, estradiol (E2)<110pmol/L (or <30pg/mL) as well;
3. ≤65 years old, with no restricted activity.

Exclusion Criteria:

1. Known hypersensitivity to similar medicines or other products derived from mammalian cells, or medical history of severe allergic to foods or medicines;
2. Treatment with diphosphonate or fluoride, oestrogen, selective estrogen receptor modulators, calcitonin, parathyroid hormone, high dose Vitamin D (≥1000 IU/day), anabolic steroids, systemic glucocorticoids within 12-month before dosing, or administered with calcitriol within 6 months before dosing;
3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2.0 times the upper limit of normal (ULN), or alkaline phosphatase (ALP)>1.5×ULN, or Total bilirubin (TBIL) >1.5×ULN, creatinine clearance rate<60 mL/min;
4. Disorders that could affect the study outcomes, such as osteomalacia, dysostosis, Paget's disease, Cushing syndrome, hyperprolactinemia, rheumatoid arthritis, hyperparathyroidism, hypoparathyroidism, or other diseases that could affect bone metabolism;
5. Hyperthyroidism or hypothyroidism, unless hypothyroidism patients are receiving regular treatment with thyroid hormone and:

   * Thyroid stimulating hormone (TSH) is normal, or
   * TSH>4.78μIU/Ml, ≤10.0μIU/mL and thyroxine (T4) is normal.
6. Malabsorption syndrome or other disorders that could affect intestinal absorption function, such as Crohn's disease, chronic pancreatitis, etc;
7. Hepatocirrhosis or severe liver disease (defined as ascites, hepatic encepalopathy, coagulation disorder, hypoalbuminemia, Esophagus and fundus gastricus varication, persistent jaundice), known diseases of biliary tract (excluding Gilbert syndrome and Asymptomatic gallstone);
8. Past or currently suffering from mandibular osteomyelitis or osteonecrosis, or any fracture within 6 months prior to first dosing; or suffering from acute tooth or mandibular disease that require tooth extracting, dental implanting or other invasive surgery; or had the above operation within 1-month before first dosing; or unhealing wound of oral surgery;
9. HBsAg positive, or anti-HCV antibody positive, or anti-HIV antibody positive, or anti-Syphilis antibody positive;
10. Prior malignancies (excluding the targeted breast cancer, basal cell carcinoma, or cervical cancer in situ) within 5 years (excluding completely resected Basal cell or squamous-cell carcinoma in situ, cervical carcinoma and Breast ductal carcinoma；
11. A variety of diseases that affect the ability of the subject to sign informed consent or follow the steps of the study; or suffer from various physical or mental illnesses that the investigators consider to affect the subject's successful completion of the study or may interfere with the interpretation of the findings;
12. Albumin-adjusted calcium≥2.0mmol/L, ≤2.9mmol/ L(Calcium supplements are not allowed within 8 hours before examination);
13. Subjects with fracture high risk and requiring treatment;
14. Has been selected for the study of other test devices or test drugs, or the duration of the clinical studies that have taken less than 30 days or 5 half-lives or biological effects, whichever is longer.
15. Other situations which are not suitable for participation judged by the principal investigator (PI).

Max Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events （AEs） | Up to 252 days.
  Include physical findings, changes in laboratory values, vital signs, and 12-lead electrocardiogram (ECG) data.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to time 'last' where last is the last time point after administration [AUClast] | Up to 252 days.
  Calculated by the linear trapezoidal method.
Area under the plasma concentration-time curve from time zero to infinity [AUC0-inf] | Up to 252 days.
  Calculated by the linear trapezoidal and extrapolation method.
Maximum observed maximum plasma concentration [Cmax] | Up to 252 days.
  The maximum (or peak) serum concentration that TK006 achieves after the drug has been administrated and before the administration of a second dose.
Time to reach the maximum observed plasma concentration [Tmax] | Up to 252 days.
  The time at which the Cmax is observed.
Terminal elimination half-life[T1/2] | Up to 252 days.
  The time required to divide the plasma concentration by two after reaching pseudo-equilibrium, and not the time required to eliminate half the administered dose.
Bioavailability corrected apparent volume of the central compartment cleared of drug per unit [Cl/F] | Up to 252 days.
  The apparent volume of the central compartment cleared of drug per unit time was estimated using the formula: Cl/F = Dose / AUC0-∞
Bioavailability corrected apparent volume of distribution [Vd/F] | Up to 252 days.
  Apparent volume of distribution based on the terminal elimination phase.
Serum type I collagen cross-link C telopeptide (sNTX) | Up to 252 days.
  Would be assessed at day1, 3, week 1, 2, 4, 8, 12, 16, 20, 24, 28, 32 and 36.
serum bone alkaline phosphatase [bALP] | Up to 252 days.
  Would be assessed at week 1, 2, 4, 8, 12, 16, 20, 24, 28, 32 and 36.
Intact Parathyroid Hormone (iPTH) | Up to 252 days.
  Would be assessed at day1, 3, week 1, 2, 4, 8, 12, 16, 20, 24, 28, 32 and 36.
Bone density of lumbar vertebra and collum femoris | Up to 252 days.
  Assessed by Dual energy X-ray (DXA) bone density measurement at week 8,16, 24 and 36.
anti-drug antibody [ADA] | Up to 252 days.
  Assessed at day 0（pre-dosing）, week 4, 12, 24 and 36.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang H Y, Study Director — Jiangsu T-Mab Biopharma Co.,Ltd
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China